Lifebox Project IRAS No: 211895



Great Ormond Street London WC1N 3JH T: +44 (0)20 7405 9200

## Development of a robust and reliable pulse oximeter for use by frontline healthcare providers caring for children with pneumonia in low-income countries CONSENT FORM

This study (Project ID: 15HC31) has been given favourable review for conduct in the NHS by: XXXX Research Ethics Committee on date YYYY

Please initial all boxes

| 1. | I confirm that I have read and understand the information sheet dated XXX (version 1.0) for the above study. I have had the opportunity to consider the information and ask questions and I have had my questions answered satisfactorily. | | |
|---|---|---|---|
| 2. | 7 1 1 | y participation is voluntary and that I am free to withdraw consent to participate at iving any reason, without my legal rights being affected. | |
| 3. | I understand that my views may be audio-recorded and I consent to the use of this material by the research team, possibly including verbatim quotes. | | |
| 4. | I understand that information provided for this study will be treated as strictly confidential and handled in accordance with the Data Protection Act 1998. I am assured that no personal identifying information will be kept which could link me to any data recorded. | | |
| 5. | I understand that data collected during the study may be looked at by individuals from Great Ormond Street Hospital, or from regulatory authorities. | | |
| 6. | I consent to take part in this study | | |
| Name of healthcare worker | | Date | Signature |
| Name of person taking consent | | Date | Signature |

You will be given a copy of this information sheet and signed consent form for your records.

Thank you for your time.

Healthcare worker consent Date of issue: 24<sup>th</sup> October 2016 Consent form version number: v1